CLINICAL TRIAL: NCT04418050
Title: Prosthetic Arthroplasties in Weight-bearing Shoulders in Individuals With Long-term Wheelchair Use
Brief Title: Prosthetic Arthroplasties in Weight-bearing Shoulders
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0200
Record Dates: First submitted 2020-04-17; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-03

CONDITIONS: Prosthetic Arthroplasties
Keywords: paraplegia; Shoulder prosthesis; spinal cord injury; wheelchair
MeSH Terms: conditions — Paraplegia; Spinal Cord Injuries | interventions — Arthroplasty, Replacement, Shoulder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Shoulder arthroplasty — Surgery consisting in replacement of gleno-humeral joint by a shoulder prosthesis

SUMMARY:
Repeated transfers and wheelchair propulsion in patients with neurological deficit of the lower limbs leads to a major mechanical overload of the upper limbs, especially on shoulders, the "weight-bearing" shoulder. Under these conditions, arthroplasty is subject to significant constraints; such an indication in this condition is always discussed. The objective of this study was to evaluate the medium-term clinical and functional outcomes of anatomical and reverse arthroplasty on the weight-bearing shoulder in individuals with long-term wheelchair use.

ELIGIBILITY:
Inclusion criteria:

* patients not walking or rarely walking, long-term users of a wheelchair before the intervention, and surgery on at least one shoulder by anatomical or reverse prosthesis

Exclusion criteria:

* Patient walking without aid
* Shoulder surgery other than arthroplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients not walking or rarely walking, long-term users of a wheelchair
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2010-02-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Evolution of joint mobility | 1 day
  Evolution of joint mobility

SECONDARY OUTCOMES:
number of searches for early implant loosening | 1 day
  number of searches for early implant loosening

CONTACTS AND LOCATIONS:
Overall Officials: Léo Chiche, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC